CLINICAL TRIAL: NCT02884882
Title: Emotions Analysis in Patients With Chronic Phase of Stroke Basal Ganglia: Neuropsychological and Neurophysiological Study of Changes in Emotional Experiences
Brief Title: Emotions Analysis in Patients With Chronic Phase of Stroke Basal Ganglia
Acronym: KALISS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty to recrut
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KALISS RB10.077
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Stroke Basal Ganglia
Keywords: Stroke Basal Ganglia; Emotional change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emotional induction in stroke population (Other): Six films are presented, each after a relaxation period after which the basal score is measured.
  Interventions: Other: Emotional induction
- Emotional induction in healthy volunteers (Placebo Comparator): Six films are presented, each after a relaxation period after which the basal score is measured.
  Interventions: Other: Emotional induction

INTERVENTIONS:
Other: Emotional induction — Score (from 1 to 10) rated the felt for each target emotions for the following 6 dimensions: joy, sadness, fear, disgust, anger, no emotion, after the presentation of short sequences of standardized films.

SUMMARY:
Compare the emotional experience of patients with focal lesions of the basal ganglia by ischemic or hemorrhagic damage and healthy participants. These anomalies will be highlighted by neuropsychological and electrophysiological assessments.

ELIGIBILITY:
Inclusion Criteria:

* For cases :

  * right-handed patient
  * ischemic or hemorrhagic stroke older than 3 months with single lesion preferably less than 20 mm in diameter affecting the basal ganglia and sparing cortex
  * Rankin score estimated prior stroke must be equal to 0 and after stroke <3 (at inclusion).
* For participants control : right-handed patient

Exclusion Criteria:

* For cases : severe aphasia - Prosopagnosia apperceptive - cerebral neurological pathology associated history, especially dementia - History of depression and psychiatric disorders treated - another stroke vascular territory than that for which the patient is included - diffuse lesions of the white matter Fazekas a score of> 2 (periventricular or subcortical) - Contraindications to MRI
* For participants control : No history neurosurgical - No history of head trauma with loss of consciousness - not known neurological disease - not known psychiatric illness - No psychotropic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The emotional experience | Baseline
  The emotional response will be compared between patients with focal lesion cores by ischemic or hemorrhagic reached that of healthy participants.
  Score (from 1 to 10) rated the felt for each target emotions for the following 6 dimensions: joy, sadness, fear, disgust, anger, no emotion, after the presentation of short sequences of standardized films. Six films are presented, each after a relaxation period after which the basal score is measured.

SECONDARY OUTCOMES:
The recognition of facial expressions | Baseline
  The facial expression recognition will be compared between patients with focal lesion cores by ischemic or hemorrhagic reached that of healthy participants.
  Percentage of recognition of facial emotions expression for each of the following 7 sizes: joy, sadness, fear, surprise, disgust, anger, no emotion; 8 frames per dimensions are presented on a total of 56 facial expressions (Ekman & Friesen, and Karolinska series).

CONTACTS AND LOCATIONS:
Overall Officials: Serge TIMSIT, Principal Investigator — Centre Hospitalier Régional de Brest
Locations (1):
- Centre Hospitalier Régional Universitaire de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No